CLINICAL TRIAL: NCT03974295
Title: The Impact of Vaginal Intercourse on Pregnancy Rates After Frozen Embryo Transfer; A Single Blinded Randomized Trial.
Brief Title: The Impact of Vaginal Intercourse on Pregnancy Rates After Frozen Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00040515
Record Dates: First submitted 2019-05-20; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Infertility; Pregnancy Related; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: After informed consent signing and randomization using a computer generated randomization scheme, the Research Nurse will open a numbered, opaque, and sealed envelope, within which there will be a white sheet of paper labelled with the patient assigned group. The participant will be informed of their assigned group by the Research Nurse. Patients assigned to the study group will be handed a log to record the number of times the patient engages in unprotected vaginal intercourse. The fertility providers will be blinded to the patients assigned treatment group. Patients who do not consent to be part of the study will still undergo their planned frozen embryo transfer per protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercourse Group (Experimental): unlimited unprotected vaginal intercourse starting 24 hours after the frozen embryo transfer
  Interventions: Behavioral: Vaginal unprotected intercourse
- Pelvic Rest Group (No Intervention): pelvic rest after frozen embryo transfer until positive pregnancy test

INTERVENTIONS:
Behavioral: Vaginal unprotected intercourse — Patients will allowed to engage in vaginal unprotected intercourse as many times as desired after 24 hours of pelvic rest after a frozen embryo transfer.
  Arms: Intercourse Group

SUMMARY:
This study aims to evaluate whether allowing unprotected vaginal intercourse 24 hours after frozen embryo transfer will result in higher ongoing clinical pregnancy rates in comparison to having participants abstain from unprotected vaginal intercourse until pregnancy test (10-14 days after frozen embryo transfer).

DETAILED DESCRIPTION:
Given the overwhelming evidence suggesting beneficial effect of seminal plasma on embryo implantation, we sought to explore this benefits in in vitro fertilization treatments by limiting the study cohort to those having frozen embryo transfer with programmed hormone replacement for endometrial preparation and some form of parenteral progesterone supplementation. This design will enable us to overcome the concerns and limitations of all previous studies. In this study, patients will be randomized into two groups, group 1 will have their frozen embryo transfer followed by current standard of care (no unprotected vaginal intercourse until pregnancy test) and group 2 will have their frozen embryo transfer followed by unlimited unprotected vaginal intercourse starting 24 hours after transfer. The primary endpoint of the study will be ongoing clinical pregnancy

rates in the two groups while secondary endpoints will include implantation, positive pregnancy, miscarriage and live birth rates. Overall, this study aims to investigate whether the elimination of current universal pelvic rest protocol in patients undergoing frozen embryo transfer will help optimize pregnancy outcomes.

This study aims to evaluate whether allowing unprotected vaginal intercourse 24 hours after frozen embryo transfer will result in higher ongoing clinical pregnancy rates in comparison to having participants abstain from unprotected vaginal intercourse until pregnancy test (10-14 days after frozen embryo transfer).

ELIGIBILITY:
Inclusion Criteria:

* female fertility patients having frozen embryo transfer
* programmed hormone replacement (Oral Estrace, Vivelle dot (patch), intravenous Estradiol) with and without gonadotrophin releasing hormone analogue pretreatment and some form of parenteral progesterone supplementation (daily or every 3 days intramuscular Progesterone) for luteal support

Exclusion Criteria:

* unable to provide informed consent
* not undergoing programmed hormone replacement for frozen embryo transfer (natural cycle frozen embryo transfer)
* undergoing fresh embryo transfer
* not able to engage in heterosexual intercourse (same sex couple, partner with severe sexual dysfunction)
* cannot undergo unprotected vaginal intercourse (infected with hepatitis B, C, or human immunodeficiency virus).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only patients undergoing embryo transfer will be candidates for the study.
Enrollment: 400 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rates | up to 2 years
  A serum quantitative pregnancy test will be performed 10-14 days following the frozen embryo transfer per clinic protocol. Positive pregnancy test is defined a serum quantitative beta hCG > 5 mU/mL.

SECONDARY OUTCOMES:
Implantation rates | up to 2 years
  Implantation rate will be defined as number of gestational sacs observed at echographic screening at 6 weeks of pregnancy divided by the number of embryos transferred.
Clinical pregnancy rate | up to 2 years
  Ongoing clinical pregnancy rate is defined as presence of a fetal heartbeat at 6-7 weeks of pregnancy.
Biochemical pregnancy rate | up to 2 years
  Biochemical pregnancy rate is defined as positive pregnancy test or elevated β-hCG level which does not result in implantation.
Miscarriage rate | up to 2 years
  Miscarriage rate is defined as a pregnancy loss is the loss of a fetus that occurs before 20 weeks of gestation.
Live birth rate | up to 2 years
  Live birth rate is defined as number of deliveries that resulted in a live born neonate, expressed per 100 embryo transfers.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gaikwad S, Garrido N, Cobo A, Pellicer A, Remohi J. Bed rest after embryo transfer negatively affects in vitro fertilization: a randomized controlled clinical trial. Fertil Steril. 2013 Sep;100(3):729-35. doi: 10.1016/j.fertnstert.2013.05.011. Epub 2013 Jun 10. PMID 23755954
- [Background] Lambers MJ, Lambalk CB, Schats R, Hompes PG. Ultrasonographic evidence that bedrest after embryo transfer is useless. Gynecol Obstet Invest. 2009;68(2):122-6. doi: 10.1159/000226283. Epub 2009 Jul 3. PMID 19590224
- [Background] Su TJ, Chen YC, Hung YT, Yang YS. Comparative study of daily activities of pregnant and non-pregnant women after in vitro fertilization and embryo transfer. J Formos Med Assoc. 2001 Apr;100(4):262-8. PMID 11393126
- [Background] Li B, Zhou H, Li W. Bed rest after embryo transfer. Eur J Obstet Gynecol Reprod Biol. 2011 Apr;155(2):125-8. doi: 10.1016/j.ejogrb.2010.12.003. PMID 21300426
- [Background] Purcell KJ, Schembri M, Telles TL, Fujimoto VY, Cedars MI. Bed rest after embryo transfer: a randomized controlled trial. Fertil Steril. 2007 Jun;87(6):1322-6. doi: 10.1016/j.fertnstert.2006.11.060. Epub 2007 Mar 23. PMID 17362946
- [Background] Botta G, Grudzinskas G. Is a prolonged bed rest following embryo transfer useful? Hum Reprod. 1997 Nov;12(11):2489-92. doi: 10.1093/humrep/12.11.2489. PMID 9436691
- [Background] Sharif K, Afnan M, Lenton W, Khalaf Y, Ebbiary N, Bilalis D, Morgan C. Do patients need to remain in bed following embryo transfer? The Birmingham experience of 103 in-vitro fertilization cycles with no bed rest following embryo transfer. Hum Reprod. 1995 Jun;10(6):1427-9. doi: 10.1093/humrep/10.6.1427. PMID 7593509
- [Background] Rezabek K, Koryntova D, Zivny J. [Does bedrest after embryo transfer cause a worse outcome in in vitro fertilization?]. Ceska Gynekol. 2001 May;66(3):175-8. Czech. PMID 11464374
- [Background] Aoki Y, Kumakiri J, Itakura A, Kikuchi I, Takahashi N, Satoru T. Should sexual intercourse be avoided during the embryo transfer cycle? Life-threatening ruptured heterotopic pregnancy after single thawed embryo transfer: case report and review of the literature. Clin Exp Obstet Gynecol. 2017;44(3):489-491. PMID 29949304
- [Background] Schjenken JE, Robertson SA. Seminal Fluid Signalling in the Female Reproductive Tract: Implications for Reproductive Success and Offspring Health. Adv Exp Med Biol. 2015;868:127-58. doi: 10.1007/978-3-319-18881-2_6. PMID 26178848
- [Background] Gutsche S, von Wolff M, Strowitzki T, Thaler CJ. Seminal plasma induces mRNA expression of IL-1beta, IL-6 and LIF in endometrial epithelial cells in vitro. Mol Hum Reprod. 2003 Dec;9(12):785-91. doi: 10.1093/molehr/gag095. PMID 14614040
- [Background] Sharkey DJ, Macpherson AM, Tremellen KP, Mottershead DG, Gilchrist RB, Robertson SA. TGF-beta mediates proinflammatory seminal fluid signaling in human cervical epithelial cells. J Immunol. 2012 Jul 15;189(2):1024-35. doi: 10.4049/jimmunol.1200005. Epub 2012 Jun 15. PMID 22706080
- [Background] Laird SM, Tuckerman EM, Dalton CF, Dunphy BC, Li TC, Zhang X. The production of leukaemia inhibitory factor by human endometrium: presence in uterine flushings and production by cells in culture. Hum Reprod. 1997 Mar;12(3):569-74. doi: 10.1093/humrep/12.3.569. PMID 9130761
- [Background] Lim KJ, Odukoya OA, Ajjan RA, Li TC, Weetman AP, Cooke ID. The role of T-helper cytokines in human reproduction. Fertil Steril. 2000 Jan;73(1):136-42. doi: 10.1016/s0015-0282(99)00457-4. PMID 10632428
- [Background] von Wolff M, Thaler CJ, Strowitzki T, Broome J, Stolz W, Tabibzadeh S. Regulated expression of cytokines in human endometrium throughout the menstrual cycle: dysregulation in habitual abortion. Mol Hum Reprod. 2000 Jul;6(7):627-34. doi: 10.1093/molehr/6.7.627. PMID 10871650
- [Background] Tremellen KP, Valbuena D, Landeras J, Ballesteros A, Martinez J, Mendoza S, Norman RJ, Robertson SA, Simon C. The effect of intercourse on pregnancy rates during assisted human reproduction. Hum Reprod. 2000 Dec;15(12):2653-8. doi: 10.1093/humrep/15.12.2653. PMID 11098040
- [Background] Crawford G, Ray A, Gudi A, Shah A, Homburg R. The role of seminal plasma for improved outcomes during in vitro fertilization treatment: review of the literature and meta-analysis. Hum Reprod Update. 2015 Mar-Apr;21(2):275-84. doi: 10.1093/humupd/dmu052. Epub 2014 Oct 3. PMID 25281684
- [Background] Nawroth F, von Wolff M. Seminal Plasma Activity to Improve Implantation in In Vitro Fertilization-How Can It Be Used in Daily Practice? Front Endocrinol (Lausanne). 2018 Apr 27;9:208. doi: 10.3389/fendo.2018.00208. eCollection 2018. No abstract available. PMID 29755413
- [Background] Steiner AZ, Pritchard DA, Young SL, Herring AH. Peri-implantation intercourse lowers fecundability. Fertil Steril. 2014 Jul;102(1):178-82. doi: 10.1016/j.fertnstert.2014.03.017. Epub 2014 Apr 18. PMID 24746744
- [Background] von Wolff M, Rosner S, Germeyer A, Jauckus J, Griesinger G, Strowitzki T. Intrauterine instillation of diluted seminal plasma at oocyte pick-up does not increase the IVF pregnancy rate: a double-blind, placebo controlled, randomized study. Hum Reprod. 2013 Dec;28(12):3247-52. doi: 10.1093/humrep/det351. Epub 2013 Sep 17. PMID 24045780